CLINICAL TRIAL: NCT05512247
Title: Use of Home-delivered Meals to Manage Cardiometabolic Health During Pregnancy Among Predominantly Black, Low-income Women in Alabama
Brief Title: Hearty Meals for Mom- Pilot Study of Meal Delivery for Cardiometabolic Health During Pregnancy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Camille S Worthington, PhD, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300009764; P50MD017338 (NIH)
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Diet, Healthy; Pregnancy
Keywords: Meal Delivery; Maternal Overweight or Obesity; Blood Pressure; Food Security; Pregnancy; Gestational Weight Gain
MeSH Terms: conditions — Obesity; Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: All participants will receive the meal delivery intervention to examine feasibility metrics (e.g., recruitment, attrition, adherence, safety) and pre-post intervention changes. A quasi-experimental design utilizing a comparison group derived from de-identified hospital records will be used for exploratory analyses of intervention impact on gestational weight gain and blood pressure compared to standard care.
Masking Description: All participants enrolled in the study will receive the meal delivery intervention, so blinding is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal Delivery (Experimental): Behavioral intervention program designed to improve diet quality and promote healthy weight gain in women with overweight/obesity through meal delivery and behavioral strategies during pregnancy.
  Interventions: Behavioral: Meal Delivery

INTERVENTIONS:
Behavioral: Meal Delivery — 10 home-delivered meals per week provided by a local meal delivery company + brief weekly behavioral support with study staff

SUMMARY:
This study is being done to assess the feasibility, acceptability, and preliminary impact of a meal delivery intervention designed to improve diet quality and promote appropriate gestational weight gain among predominantly Black and low-income pregnant women with overweight or obesity. This will be done by 1) assessing the feasibility and acceptability of the meal delivery intervention; 2) investigating changes in patient-reported diet quality, barriers to healthy eating, and food security; and 3) exploring the preliminary impact of the meal delivery intervention on gestational weight gain and blood pressure and estimate the effect size of the intervention relative to a de-identified non-randomized control group that will be derived from de-identified hospital records.

DETAILED DESCRIPTION:
Subjects will receive 10 home-delivered meals per week from about 20 weeks gestation until 40 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid eligible and/or have a household income at or below 185 percent of the federal poverty line
* 18 years of age or older
* <= 19 weeks gestation
* Currently experiencing a singleton pregnancy
* Receiving prenatal care at a University of Alabama at Birmingham clinic
* Planning to deliver at the University of Alabama at Birmingham
* Residing within the meal company's delivery radius
* Body mass index >= 25
* Willing to consent

Exclusion Criteria:

* Self-reported major health condition (such as renal disease, cancer, or Type 1 or Type 2 diabetes)
* Current treatment for severe psychiatric disorder (such as schizophrenia)
* Current substance abuse
* Self-reported diagnosis of anorexia or bulimia
* Known fetal anomaly
* Current use of medication expected to significantly impact body weight
* Planned termination of the current pregnancy
* Participation in another dietary and/or weight management intervention during the current pregnancy
* Unwilling or unable to understand and communicate in English
* Unwilling or unable to consume study meals

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Healthy Eating Index score from baseline to follow-up | three 24-hour dietary recalls on non-consecutive days at baseline (18-22 weeks gestation) and follow-up (33-37 weeks gestation)
  Determined based on the Healthy Index Score, in which 100 indicates complete alignment with the Dietary Guidelines for Americans and 0 is the minimum score, as calculated from three 24-hour dietary recalls conducted on non-consecutive days (2 weekdays + 1 weekend day) at each time point.

SECONDARY OUTCOMES:
Change in Food Security | baseline (18-22 weeks gestation), (33-37 weeks gestation)
  Determined using the 18-item United States (US) Household Food Security Survey Module based on the previous 30 days. Adult food security scores range from 0 to 10, with lower values indicating greater food security.
Change in Barriers to Healthy Eating | baseline (18-22 weeks gestation), follow-up (33-37 weeks gestation)
  Participants will be asked to score 5 statements corresponding to different barriers to healthy eating on a 5-point Likert scale ranging from strongly agree to strongly disagree (adapted from Sibai D et al. 2022). Changes in the distribution of responses to each barrier will be assessed, as well as changes in the proportion of women somewhat/strongly agreeing with each barrier will be compared.
Study Participation Rate | baseline (18-22 weeks gestation)
  Percentage of eligible subjects who agreed to participate out of those who were screened.
Participant Retention | baseline (18-22 weeks gestation), follow-up (33-37 weeks gestation)
  The proportion of enrolled participants who complete follow-up
Participant Adherence to Intervention | Collected weekly from intervention start (20-24 weeks gestation) to intervention end (40 weeks gestation)
  Proportion of weekly study meals participants consumed based on responses to weekly electronic surveys in which participants will report the number of study meals a) they consumed, b) other household members consumed, or c) that were uneaten.
Change in Participant Satisfaction with Diet | baseline (18-22 weeks gestation), follow-up (33-37 weeks gestation)
  To assess satisfaction with the study intervention, the 28-item Diet Satisfaction Questionnaire will be used in which participants respond to 28 statements using a 5-point Likert scale. Responses are average to produce a total diet satisfaction score ranging from 1-5. Changes in overall diet satisfaction, as well as changes in subscale scores for Cost Factor and Planning & Preparation Factor will be examined from baseline to follow-up.

OTHER OUTCOMES:
Change in Blood Pressure | First prenatal visit through delivery (Collected once at study end from medical record)
  Systolic and diastolic blood pressure measured at each prenatal visit will be retrieved from medical records for all participants at the end of the intervention.
Gestational weight gain | First prenatal visit through delivery (Collected once at study end from medical record)
  Weight measured at each prenatal visit will be retrieved from medical records for all participants at the end of the intervention and used to calculate total gestational weight gain and rate of gestational weight gain.

CONTACTS AND LOCATIONS:
Overall Officials: Camille S Worthington, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in a publication will be made available upon request beginning 9 months and ending 36 months following article publication. The research team will keep a record of all individuals and/or research teams who request and receive a copy of the project data. Interested investigators will be asked to submit a document indicating the specific aims of the analyses, the analytic plan, available resources for completing the proposed project, proposed timeline, and goals (i.e., manuscripts, presentations, and/or grant applications). The PI and research team will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to complete the request, and whether data will be adequately protected and managed.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after publication of results and ending 36 months following article publication.
Access Criteria: Access to IPD stripped of all HIPAA identifiers (except age) for this study can be requested by qualified researchers engaging in independent scientific research whose proposed research has received Institutional Review Board approval, and will be provided following review and approval of a research proposal and timeline, statistical analysis plan, and goals (e.g., manuscripts, presentations, grant applications). The Principal Investigator (PI) and research team will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to complete the request, and whether data will be adequately protected and managed. Based on institutional policies, execution of a Data Sharing Agreement may be required prior to sharing of IPD. IPD requests can be made to the PI at cschneid@uab.edu.